CLINICAL TRIAL: NCT03108053
Title: Results of a Prospective Randomized Trial of Safety Guidewire Use in Ureteroscopic Stone Surgery: to Use or Not to Use
Brief Title: Results of Safety Guidewire Use in Ureteroscopic Stone Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAR.UAD.001; 09.2017.098 (Other: Clinical Research Ethics Committee of Marmara University)
Record Dates: First submitted 2017-03-10; First posted 2017-04-11 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Urinary Stone
Keywords: urinary stones; semirigid ureteroscopy; guidewire
MeSH Terms: conditions — Urinary Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guidewire used (Active Comparator): Patients whose semirigid ureteroscopy procedure is conducted with the use of safety guidewire
  Interventions: Procedure: Semirigid Ureteroscopy (URS) With Guide Wire
- No guide wire used (Experimental): Patients whose semirigid ureteroscopy procedure is conducted without the use of safety guidewire
  Interventions: Device: Semirigid Ureteroscopy (URS) Without Guide Wire

INTERVENTIONS:
Procedure: Semirigid Ureteroscopy (URS) With Guide Wire — Semirigid URS is the operations used for ureteral stone disease. In routine practice it is most commonly done with the use of a guide wire. It is conducted with ureteroscope and stone is disintegrated most commonly with lasers.
  Arms: Guidewire used
Device: Semirigid Ureteroscopy (URS) Without Guide Wire — Semirigid URS is the operations used for ureteral stone disease . It is conducted with ureteroscope and stone is disintegrated most commonly with lasers.
  Arms: No guide wire used

SUMMARY:
Up-to-date, urology guidelines introduce safety guidewire (SGW) as an integral tool in ureteroscopy and recommended its routine use. However, the necessity of SGW placement in endourological procedures lack evidence and is being suggested as an expert opinion. Present study aimed to evaluate the use of SGW placement and its necessity in treatment of ureteral stones with semi-rigid ureteroscopy (s-URS).

For this purpose patients with ureteral stones are being stratified according to ureteral stone location and prospectively randomized into two groups' according to SGW usage or not in s-URS. Ureteroscopy and litotripsy is being done with a semi-rigid ureteroscope of 6.4/7.8 Fr (Olympus) and laser. Chi-square and student t-test were used for comparing data.

ELIGIBILITY:
Inclusion Criteria:

* Ureteral stone disease patients who would undergo ureteroscopy procedure

Exclusion Criteria:

* Patients who have a medical condition that makes randomisation not possible
* Patients in whose operations safety guidewire is regarded as a necessity
* Patients who refuse to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2014-06-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Stone free rates | Post operative 3 months (12 weeks after surgery)

SECONDARY OUTCOMES:
Operation duration of surgery | the duration of surgical procedure
Late Complication rate | Post operative 3 months (12 weeks after surgery)
Early Complication rate | Post operative 3 days (up to 3 days after surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No